CLINICAL TRIAL: NCT07211243
Title: Multicenter, Randomised in Parallel Groups, Controlled Study to Compare Performance and Safety of Suprasorb®X+PHMB Pro With Suprasorb® X+PHMB Dressing in Treatment of Infected Venous Leg Ulcers
Brief Title: Suprasorb®X+PHMB Pro vs Suprasorb®X+PHMB in Treatment of Infected Venous Leg Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lohmann & Rauscher (Industry)
Collaborators: AXCELLANT (Unknown); Clean Data Labs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-07
Record Dates: First submitted 2025-09-11; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Venous Leg Ulcer
Keywords: maceration; bacterial cellulose dressing; PHMB; antimicrobial dressing
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to Suprasorb®X+PHMB Pro or Suprasorb®X+PHMB in a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: Primary endpoint ans some secondary endpoints will be re-confirmed by a blinded assessment of the wound photographs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprasorb®X+PHMB Pro (Experimental): Patients will receive the assigned wound dressing for 21 (±2) days, or till the complete epithelialization, if it occurs earlier. The patients should also receive adequate compression and, if necessary, systemic antimicrobial drug therapy.
  Interventions: Device: PHMB-impregnated biocellulose wound dressing with additional polyethylene film on top, compression therapy, systemic antomicrobial therapy (optional)
- Suprasorb®X+PHMB (Active Comparator): Patients will receive the assigned wound dressing for 21 (±2) days, or till the complete epithelialization, if it occurs earlier. The patients should also receive adequate compression and, if necessary, systemic antimicrobial drug therapy.
  Interventions: Device: PHMB-impregnated biocellulose wound dressing without additional polyethylene film on top, compression therapy, systemic antomicrobial therapy (optional)

INTERVENTIONS:
Device: PHMB-impregnated biocellulose wound dressing with additional polyethylene film on top, compression therapy, systemic antomicrobial therapy (optional) — Application of a wound dressing with additional polyethylene film on top and compression therapy. Optional usage of the systemic antimicrobial therapy.
  Arms: Suprasorb®X+PHMB Pro
Device: PHMB-impregnated biocellulose wound dressing without additional polyethylene film on top, compression therapy, systemic antomicrobial therapy (optional) — Application of a wound dressing without additional polyethylene film on top and compression therapy. Optional usage of the systemic antimicrobial therapy.
  Arms: Suprasorb®X+PHMB

SUMMARY:
This clinical investigation will be conducted as a multicentre, open-label, randomised in parallel groups, controlled study on patients with infected venous leg ulcers.

DETAILED DESCRIPTION:
During the screening, all patients will be assessed for inclusion and exclusion criteria and wound exudation status. Eligible patients with slight or moderate wound exudation will be randomly assigned to treatment with either Suprasorb®X+PHMB Pro or Suprasorb®X+PHMB. The patients who fulfil all other eligibility criteria but have high level of wound exudation will enter a 7-days run-in period, during which they will receive superabsorbent dressing (e.g. Vliwazell® Pro, Vliwasorb® Pro) and monitored compression therapy with Rosidal® 1C. During the run-in period they should receive appropriate treatment including systemic antimicrobial drug therapy if required. After this time, these patients should be re-assessed and in case they still fulfil all eligibility criteria, and the exudation decreased at least to a moderate level, they will be randomised to Suprasorb®X+PHMB Pro or Suprasorb®X+PHMB. In case the exudation would not decrease within this period or other eligibility criteria are not met anymore, they will be screened out.

Upon randomisation, all patients will receive the assigned dressing for 21 (±2) days, or till the complete epithelialization, if it occurs earlier. The patients should also continue to receive adequate compression and, if necessary, systemic antimicrobial drug therapy. During the study participation, selected parameters of the wound will be assessed at Baseline, Interim Visit, and EOT visit. In addition, dressing changes may be performed in-between on as needed basis. After 3 weeks of treatment with Suprasorb®X+PHMB Pro or Suprasorb®X+PHMB, all patients will complete the study. Their further treatment (if necessary), will not be the part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Infected* venous** leg ulcer
* Slightly to moderately exuding wound***
* Patient has signed informed consent

  * as per CDC definition, also TILI score ≥ 5 ** ABPI > 0.8 and < 1.2 *** patients with highly exuding wounds may be screened for a 7 days run-in period to receive superabsorbent dressing and monitored compression therapy and re-con-sidered for enrolment in case the exudation level decreases

Exclusion Criteria:

* Participation in other interventional clinical trial that could interfere with the present study within 4 weeks of the randomisation and during the whole duration of this study
* Wounds with exposed cartilage tissue (hyaline cartilage)
* Contraindications to compression therapy (e.g.: advanced peripheral ar-terial occlusive diseases, decompensated cardiac insufficiency, septic phlebitis, phlegmasia coerulea dolens, sensation disorders of the skin)
* Known allergy and/or hypersensitivity to any components of the study product or concomitant products (e.g. compression bandage)
* Any other medical condition, which, by opinion of the investigator, may have impact of the success of the study treatment and / or interpreta-tion of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Rate and severity of maceration after 3 weeks of treatment with Suprasorb®X+PHMB (Pro) | 3 weeks
  on a 4-grade scale there 0 means no maceration and 4 means severe maceration

SECONDARY OUTCOMES:
Wound area change over time | 3 weeks
  in mm2
Change of necrotic & fibrinous & granulation tissue rate in the wound bed | 3 weeks
  in %
Change of wound infection status | 3 weeks
  by a TILI (Therapeutical Index for Local Infections) score with a range 1-6. TILI < 5 indicates a wound without infection, whereas TILI ≥ 5 means a local wound infection.
Product safety (rate of product-related complications) | 3 weeks
  by rate of product-related complications
Change of wound exudation and presence of peri-wound oedema | 3 weeks
  by the investigators' assessment of exudation grade
Change in patient's pain | 3 weeks
  By NRS (numeric rating scale), with zero meaning "no pain" and 10 meaning "the worst pain imaginable"
Product usability | 3 weeks
  by user and patient questionnaire
Change in patient's quality of life | 3 weeks
  by Wound QoL-17 (wound quality of life) questionnaire
Oedema chamge | 3 weeks
  by measurement of limb circumference
Sub-bandage pressure levels retention | 3 weeks
  difference of the pressure levels, measured at the time of application and before the next dressing change with a wireless sensor

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Pańczak, MD, Principal Investigator — LECRAN - CENTRUM OPIEKI NAD RANAMI-KUNICKIEGO
Locations (8):
- Poland (8):
  - Centrum Medyczne Ultramed, Krakow
  - MelissaMed Poradnia Chirurgiczna, Lodz
  - Mikomed Spółka Z Ograniczoną Odpowiedzialnością, Lodz
  - Niepubliczny Zakład Opieki Zdrowotnej "Argo" Centrum Medyczne, Lodz
  - PP CLINIC Pietrzyk spółka partnerska lekarzy, Lublin
  - SPECJALISTYCZNY OSRODEK LECZNICZO BADAWCZY, Zbigniew Żęgota, Ostróda
  - Lecran - Centrum Opieki Nad Ranami-Kunickiego, Wroclaw
  - Specjalistyczna Pomoc Medyczna "Medservice", Zabrze

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT07211243/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT07211243/SAP_001.pdf